CLINICAL TRIAL: NCT05190484
Title: An International, Prospective, Observational Study of Patients With Chronic Inflammatory Diseases, to Assess 12-months Persistence Drivers After Switching to an Adalimumab Biosimilar, Idacio®, in a Real World Setting
Brief Title: bIosimilar of aDalimumab, an European evAluation
Acronym: IDEA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Other Study IDs: ADAL-004-CNI
Record Dates: First submitted 2022-01-04; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Psoriatic Arthritis; Crohn Disease; Ulcerative Colitis
Keywords: adalimumab; biosimilar
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Arthritis, Psoriatic; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study objective is aimed to describe all country, site, investigator and patient variables that lead to treatment persistence for at least 12 months among patients with rheumatologic and intestinal chronic inflammatory diseases who were switched to FK adalimumab, in order to develop a model to predict persistence at 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, male or female.
2. Patients diagnosed with one chronic inflammatory rheumatological (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis) or chronic inflammatory bowel (Crohn's disease, ulcerative colitis) diseases.
3. Patients who have been switched to FK adalimumab from the reference product (Humira®) or another adalimumab biosimilar.
4. Patients who have been prescribed FK adalimumab according to the SmPC prior to the inclusion.
5. Patients able to understand and complete the study questionnaires in local language during the study visits.
6. Patients willing to sign informed consent to meet data protection requirements

Exclusion Criteria:

1. Unwillingness to provide written informed consent.
2. Patients participating or expected to participate in any randomised clinical trial during their treatment with FK adalimumab.
3. Patients not expected to be available for study visits during 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female adult patients with an IMID who were prescribed FK adalimumab, meet all the study inclusion criteria and none of the exclusion criteria and provide written informed consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2022-04-30 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
TREATMENT DISCONTINUATION | 12 months
  A patient will be considered to have discontinued FK adalimumab (not persistent) if the investigator reports a permanent discontinuation or if the patient has been more than 90 consecutive days not covered by treatment (based on the refills reported).